CLINICAL TRIAL: NCT04725526
Title: Development and Efficiency of an mHealth Intervention on the Health Literacy Improvement and Self-management of the Multi-pathological Patient With Heart Failure: a Randomized Controlled Trial.
Brief Title: Efficiency of an mHealth Intervention on the Health Literacy Improvement and Self-management.
Acronym: PBS-MHE-2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PBS-MHE-2019
Record Dates: First submitted 2020-12-10; First posted 2021-01-26 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure; Multi-pathology
Keywords: mHealth intervention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual clinical practice (No Intervention): A group of pluripatological patients with heart failure and complex needs of health will be tratad per standard of care on site
- mHealth intervention plus usual clinical practice (Experimental): A group of pluripatological patients with heart failure and complex needs of health will be tratad per standard of care plus mHealth intervention on site
  Interventions: Device: Mobile phone compatible with iOS or Android

INTERVENTIONS:
Device: Mobile phone compatible with iOS or Android — MHealth (mobile health) intervention is an act whose purpose is to improve, maintain, promote or modify health, functioning or health conditions.
  Arms: mHealth intervention plus usual clinical practice

SUMMARY:
Multipathological patients with complex health needs are responsible for the majority number of avoidable hospital admissions.

The expansion of mHealth interventions in the field of communication with the patient, the reduction of health inequalities, the improvement in access to health resources, the adherence to treatments and self-care of chronic diseases lead to an optimistic horizon . However, there are few applications that demonstrate its effectiveness in these patients, which is diminished when they are not based on evidence, nor are designed by and for users with different levels of health literacy.

DETAILED DESCRIPTION:
Objective: to evaluate the efficacy of an mHealth intervention, with respect to routine clinical practice, to improve health literacy and self-management of the multiple pathological patient with heart failure and complex health needs.

Hypothesis: the proposed mHealth intervention is more effective than usual clinical practice, favoring health literacy and self-management of multiple pathological patients with heart failure and complex health needs, so its use would be relevant as part of the assistance process.

Methodology: randomized, controlled, multicenter clinical trial for the evaluation of the efficacy of an mHealth intervention with two groups: a control group (routine clinical practice) and an experimental group (routine clinical practice together with ad hoc designed mHealth intervention).

In this project, the design and content validation of the mHealth tool will be carried out, evaluating its relevance and suitability.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes and over 18 years of age;
* Attended by the health professionals of the Basic Health Areas that are participating in the study;
* Patients that give their consent to participate in the study by signing an informed consent;
* Patients that have a mobile device (Smartphone or Tablet) compatible with the Android or iOS operating system;
* Patients considered as multi-pathological based on the following criteria from those described in the Integrated Healthcare Process (Ollero et al., 2018):
* Be classified in clinical category A of chronic pathologies due to heart failure that, in a situation of clinical stability, has been in NYHA grade II, being able to be simultaneously classified, or not, in other clinical categories due to suffering from another disease Chronicles.
* Patients with at least one of the following complexity criteria: Extreme polypharmacy (10 or more active ingredients for chronic prescription); Socio-family risk (score on the Gijon scale greater than 10 points); Stage II or higher pressure ulcers; Malnutrition (BMI <18.5); Feeding with chronic and prescription tube (3 or more months); Two or more hospital admissions in the previous 12 months.

Exclusion Criteria:

* Patients with sensory deficits and/or mobility problems in the upper limbs that prevent them from using the application correctly, despite using the accessibility features of mobile devices;
* Patients with persistent cognitive impairment (Pfeiffer test with 5 or more errors or Lobo's mini-cognitive exam <23 points) and / or severe mental disorder;
* Patients with serious limitations for AVBD (Barthel index <20 points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Health literacy | 1 year
  Literacy on health defined by points (range 0-50)
General selfmanagement | 1 year
  Selfmanagement on health (scale 1-5)
selfmanagement on heart failure | 1 year
  European Heart Failure SelfCare Behavior Scale (range 12-60)

SECONDARY OUTCOMES:
self-independence | 1 year
  Personal grade of self-independence- Barthel Index
self-independence 2 | 1 year
  Personal grade of self-independence- Lawton and Brody Index
Adherence to treatments | 1 year
  Adherence to treatments measured by Morisky-Green Questionnaire
Prognosis | 1 year
  Life prognosis using PROFUND Index
Patient satisfaction | 1 year
  General patient satisfaction using a simple questionnarie
Patient satisfaction 2 | 1 year
  Patients satisfaction related to mHealth device

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Bas Sarmiento, MD, Principal Investigator — Instituto de investigación e innovación biomédica de Cádiz; Martina Fernández Gutiérrez, Principal Investigator — Instituto de investigación e innovación biomédica de Cádiz
Locations (2):
- Spain (2):
  - Health Management area of Gibraltar, Algeciras, Cádiz
  - F. para la Gestión de la Inv. Biomédica de Cádiz Ríos, Cadiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bas-Sarmiento P, Fernandez-Gutierrez M, Poza-Mendez M, Marin-Paz AJ, Paloma-Castro O, Romero-Sanchez JM; ASyAG_PPIC Team. Development and Effectiveness of a Mobile Health Intervention in Improving Health Literacy and Self-management of Patients With Multimorbidity and Heart Failure: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 29;11(4):e35945. doi: 10.2196/35945. PMID 35486437